CLINICAL TRIAL: NCT01466959
Title: The Effect of Citrasate Dialysate on Heparin Dose: A Randomized Cross Over Trial in Hemodialysis Patients.
Brief Title: The Effect of Citrasate Dialysate on Heparin Dose in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr Jennifer MacRae, Principal investigator, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ID24009
Record Dates: First submitted 2011-10-11; First posted 2011-11-08 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Kidney Disease
Keywords: hemodialysis; dialysate; acetate based dialysate; citrasate dialysate; heparin anticoagulation; hemodynamic stability
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AD- acetic acid dialysate (Active Comparator): AD is a standard bicarbonate based dialysate with a small amount of acetic acid which is the standard of care for dialysis.
  Interventions: Other: acetic-acid based dialysate (AD)
- CD - citrasate dialysate (Experimental): Dialysis with a citric acid based dialyasate.
  Interventions: Other: citrate dialysate (CD)

INTERVENTIONS:
Other: citrate dialysate (CD) — Citrasate (CD) is substituted as the dialysate during the patients regular dialysis run 4hours three times weekly for a period of 2 weeks. The only difference between citrasate and the regular dialysate is the lack of acetic acid.
  Other Names: Citrasate; Citric acid dialysate
  Arms: CD - citrasate dialysate
Other: acetic-acid based dialysate (AD) — Acetate based dialysate; AD is the standard dialysate used in hemodialysis runs 4 hours three times weekly. For the study it will be used for a period of 2 weeks and compared to the CD study time period.
  Other Names: Acetic acid dialysate; Acetate dialysate
  Arms: AD- acetic acid dialysate

SUMMARY:
An alternative to systemic heparin anticoagulation for HD is citrate dialysate (CD). CD contains a small amount of citric acid rather than acetic acid as the acidifying agent. The use of citrasate may lead to lower heparin requirements in hemodialysis. This is a randomized, double blinded, two-period crossover trial in HD patients to compare the effect of citrasate dialysis (CD) and usual acetic-acid based dialysate (AD) on heparin dose.

DETAILED DESCRIPTION:
The investigators will perform a randomized, double-blind, two-period crossover trial in chronic HD patients to compare the effect of citrasate dialysate (CD) and usual acetic-acid based dialysate (AD) on the cumulative intradialytic heparin dose. There is a four week run in phase followed by two weeks of intervention AD or CD followed by the remaining AD or CD intervention.

The primary outcome is change in intradialytic heparin dose achieved with citrasate compared with acetate dialysate. Secondary outcomes are the effect of CD compared with AD on systemic anticoagulation, bleeding time after HD, metabolic parameters, dialysis adequacy, inflammation, hemodynamic stability, and intra-rater and inter-rater reliability of the dialyzer clotting score.

ELIGIBILITY:
Inclusion Criteria:

* chronic stable HD patients ≥ 18 years
* on HD at least three times per week for at least 3 months

Exclusion Criteria:

* contraindication to heparin
* currently using heparin-free HD
* known clotting disorder
* on warfarin therapy
* dialyzing with a dysfunctional central venous catheter (blood flow rates consistently less than 300mL/min and/or frequent use of thrombolytic)
* history of vascular access dysfunction
* planned vascular access conversion or procedure during the study period
* use of high calcium dialysate
* active medical issue requiring hospitalization
* planned kidney transplant during the study period
* planned conversion of dialysis modality (peritoneal dialysis, nocturnal dialysis) during the study period
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The change from baseline in the cumulative dose of heparin anticoagulation used during conventional HD | 2 weeks after CD exposure, 2 weeks after AD exposure

SECONDARY OUTCOMES:
The change from baseline in the number of bleeding events, and bleeding time after HD. | After 2 weeks of exposure to CD
The change from baseline in the number of intradialytic hypotension episodes and the change from baseline in the QT interval | 2 weeks after intervention exposure
The change in small and middle solute clearance from baseline. | 2 weeks post exposure
The change from baseline on laboratory inflammatory markers as well as ionized calcium (iCa), magnesium (Mg), and bicarbonate (HCO3). | 2 weeks post exposure
The intra-rater and inter-rater reliability of our dialyzer / venous chamber clotting score. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M MacRae, MD FRCPC, Study Director — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593
- [Derived] Tai DJ, Leung K, Ravani P, Quinn RR, Scott-Douglas N, MacRae JM; Alberta Kidney Disease Network. The effect of citrate dialysate on intradialytic heparin dose in haemodialysis patients: study design of a randomised controlled trial. BMC Nephrol. 2015 Aug 25;16:147. doi: 10.1186/s12882-015-0144-z. PMID 26303208